CLINICAL TRIAL: NCT05912348
Title: The Effects of an Obesogenic Lifestyle in Recreationally Active, Young Adults
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of New Hampshire (Other)
Responsible Party: Principal Investigator, Michael Brian, Assistant Professor of Kinesiology, University of New Hampshire
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: UNH-12-FY2023_85-01
Record Dates: First submitted 2023-02-13; First posted 2023-06-22 (Actual); Last update posted 2024-07-17 (Actual); Status verified 2024-07

CONDITIONS: Insulin Resistance; Impaired Glucose Tolerance; Obesity; Metabolic Disturbance
MeSH Terms: conditions — Insulin Resistance; Glucose Intolerance; Obesity

STUDY DESIGN:
Intervention Model Description: Randomized Cross-Sectional Study Design
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Low Physical Activity and Added Carbohydrate Group (Experimental): 10-days of low physical activity (~5,000 steps/day) while consuming added sugar-sweetened beverages (~180 g/day).
  Interventions: Behavioral: Low Physical Activity and Added Carbohydrate Group
- Low Physical Activity Control (Placebo Comparator): 10-days of sedentary activity (~5,000 steps/day).
  Interventions: Behavioral: Low physical Activity Control
- Normal Activity Control (No Intervention): Maintains normal physical activity levels and exercise training
- High Physical Activity and Added Carbohydrate Group (Experimental): 10-days of high physical activity (~11,000 steps/day) while consuming added sugar-sweetened beverages (~180 g/day).
  Interventions: Behavioral: High Physical Activity and Added Carbohydrate Group

INTERVENTIONS:
Behavioral: Low Physical Activity and Added Carbohydrate Group — Young men and women will transition into a low physically active lifestyle for 10 days and consume added sugar-sweetened beverages. The intervention group will be compared to two control groups and one experimental group. One of the control groups will undergo a low physical activity intervention.
  Arms: Low Physical Activity and Added Carbohydrate Group
Behavioral: Low physical Activity Control — Young men and women will transition into a low physically active lifestyle for 10 days.
  Arms: Low Physical Activity Control
Behavioral: High Physical Activity and Added Carbohydrate Group — Young men and women will transition into a high physically active lifestyle for 10 days and consume added sugar-sweetened beverages. The intervention group will be compared to two control groups and one experimental group.
  Arms: High Physical Activity and Added Carbohydrate Group

SUMMARY:
This clinical trial aims to learn about the alterations in insulin resistance and metabolic flexibility following a transition to an obesogenic lifestyle in fit young men and women. The main questions it aims to answer are:

1. Does adding excess carbohydrates when transitioning to a sedentary lifestyle promote insulin resistance and impaired 24hr glucose regulation in healthy men and women?
2. Does adding excess carbohydrates when transitioning to a sedentary lifestyle lower the body's ability to break down fats and carbohydrates in healthy men and women?
3. Does the added physical activity blunt shifts in carbohydrate and fat oxidation in healthy men and women?

DETAILED DESCRIPTION:
Excess adiposity remains a critical health issue in the United States. Obesity and severe obesity are projected to reach approximately 34% and 9% by 2030, respectively. However, recent 2021 NHANES data reveals that our obesity and severe obesity population has already surpassed these estimates reaching 41.9% and 9.2% by 2022, respectively. While early childhood obesity has a prevalence of about 22%, which can lead to obesity during adulthood, young adulthood (20-39 years old) is another critical time where young adults without obesity or severe obesity will accumulate excess adiposity as part of this transition into middle-aged adulthood (40-59 years). In particular, young adults often transition from higher levels of physical activity (i.e., sports participation in high school, increased walking to class on college campuses, increased free time for physical activity) to lower levels of physical activity (e.g., full-time employment) and limited time to prepare healthy meals. Although obesity models tend to be complex, with multiple contributors to the development of obesity, easily accessible and rapidly digestible carbohydrates with high glycemic indexes have contributed significantly to the rise in obesity and cardiometabolic diseases in the United States.

Previous animal models have demonstrated that high carbohydrate or high-fat diets and increased sedentary activity lead to excess adiposity and insulin resistance in animal models. Animal models help us to examine mechanistic contributors to obesity and adverse cardiometabolic risks. A recently developed obesogenic lifestyle model provides an excellent model for studying the transition to an obesogenic lifestyle in healthy young adults. The obesogenic lifestyle model uses an acute exposure to a sedentary lifestyle (~5,000 steps/day) and increased carbohydrate intake (~2 liters of soda/day) for a 10-day period. Using this obesogenic lifestyle model, researchers found that the acute obesogenic lifestyle model increased insulin resistance (measured by HOMA-IR) in both men and women, but only men had declines in vascular insulin sensitivity. The reduction in vascular sensitivity is considered an early precursor for the development of metabolic dysregulation and cardiovascular disease. Nonetheless, it remains unclear whether insulin resistance and vascular insulin sensitivity were due to a lack of physical activity or increased carbohydrate intake. Further, the model must be independently validated to confirm its ability to induce insulin resistance to create a sustainable model for repeated studies.

From a behavioral aspect, the designed obesogenic lifestyle model provides an opportunity to study increases in insulin resistance when individuals transition during young adulthood into a lifestyle that induces barriers to maintaining physical activity and impairs diet quality. Importantly, this young adult population remains underrepresented in the literature compared to studies on obese or physically inactive adults. Therefore, the model has ecological relevance. The model also provides an opportunity for earlier interventions to be developed to mitigate the harmful consequences that may be offset with simple interventions that promote physical activity. Therefore, the global hypothesis of this research study is that the obesogenic lifestyle model will be a suitable model for studying the early onset of insulin resistance as it will increase insulin resistance (HOMA-IR) and impair glucose regulation in recreationally active young men and women.

ELIGIBILITY:
Inclusion Criteria:

* 18-30 years of age
* Recreationally active completing 75-150 minutes of moderate-to-vigorous intensity exercise (>2 days/week).
* Fair cardiorespiratory fitness levels (Men: VO2>38.4 ml/kg/min; Women: VO2>32.6 ml/kg/min).

Exclusion Criteria:

* Hypertension (resting or diagnosed)
* Impaired fasting blood glucose (>100mg/dL)
* Diagnosed cardiovascular disease
* Diagnosed diabetes
* Diagnosed cancer
* Diagnosed chronic kidney disease
* Diagnosed musculoskeletal disorders that prevents the individual from exercising on a bike.

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 45 (Estimated)
Dates: Start 2023-02-08 (Actual); Primary Completion 2026-09-30 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
To determine if low physical activity alone contributes to insulin resistance in healthy, recreationally active young men and women compared to men and women that reduce their physical activity and consume added sugar-sweetened beverages. | 10 days
  We will use HOMA-IR to measure changes in insulin resistance across the 4 study groups
To determine if the combined low physical activity and added carbohydrates impairs 24-hour glucose regulation compared the other study interventions. | 10 days
  Compare 24-hour glucose regulation (mmol/L) measurements across the four study groups
To determine if fat oxidation is impaired when participants reduce their physical activity levels and consume added carbohydrates compared to the three interventions | 10 days
  Compare the change in fat oxidation after the 10 day intervention

CONTACTS AND LOCATIONS:
Overall Officials: Michael S Brian, PhD, Principal Investigator — University of New Hampshire
Locations (1):
- University of New Hampshire Cardiometabolic Research Laboratory, Durham, New Hampshire, United States